CLINICAL TRIAL: NCT01589770
Title: Inflammation and the Heart
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: Arthritis Foundation (Other)
Responsible Party: Principal Investigator, C. Michael Stein, Dan May Professor of Medicine, Professor of Pharmacology, Assistant Director of the Division of Clinical Pharmacology, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 120314
Record Dates: First submitted 2012-04-24; First posted 2012-05-02 (Estimated); Results first posted 2019-04-12 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-04

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; inflammation
MeSH Terms: conditions — Arthritis, Rheumatoid; Inflammation

STUDY DESIGN:
Intervention Model Description: All participants underwent cardiac MRI(cMRI) using a 1.5 tesla Siemens Magnetom Avanto scanner to compare left ventricular structure and Left atrium size.
Who Masked: Outcomes Assessor
Masking Description: Individuals specialized in cMRI performed the analyses and were blinded to disease status of participants.
Oversight: Data Monitoring Committee: No

ARMS (2):
- rheumatoid arthritis patients (Other): People who have rheumatoid arthritis underwent cMRI
  Interventions: Other: cardiac Magnetic Resonance imaging
- controls (Other): people who do not have RA or other inflammatory disease underwent cMRI
  Interventions: Other: cardiac Magnetic Resonance imaging

INTERVENTIONS:
Other: cardiac Magnetic Resonance imaging

SUMMARY:
Studies have shown that people with rheumatoid arthritis (RA) have a higher rate of heart disease than people that do not have RA. we believe this is caused by the inflammation produced by RA.

DETAILED DESCRIPTION:
Aim 1: We want to study people with RA to see if we can detect very early changes in their heart muscle and compare these results to people who do not have RA.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age >= 18
* RA only: meet American College of Rheumatology(ACR)criteria for Diagnosis of RA
* Controls only: no evidence of RA or other inflammatory disease

Exclusion Criteria:

* Previous or current heart failure or ischemic cardiovascular disease (eg stroke, myocardial infarction, angina, CABG, stent).
* Atrial fibrillation.
* Known structural or functional cardiac abnormality, including pulmonary htn.
* Glomerular filtration rate < 60 ml/min.
* Pregnancy or breastfeeding.
* Unable to perform MRI (claustrophobia, unable to fit in magnet,pacemaker,defibrillator or non-MR safe implant).
* Hypersensitivity to gadolinium.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Michael Stein, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
all IDP that underlie results in a publication
Time Frame: 6 months after publication
Access Criteria: IPD will be shared on request made to the PI. Criteria: Data is not to be shared. Data should only be used for biomedical research. Researchers requesting access will need appropriate IRB approval and sign a data use agreement.

REFERENCES:
- [Result] Bradham W, Ormseth MJ, Elumogo C, Palanisamy S, Liu CY, Lawson MA, Soslow JH, Kawel-Boehm N, Bluemke DA, Stein CM. Absence of Fibrosis and Inflammation by Cardiac Magnetic Resonance Imaging in Rheumatoid Arthritis Patients with Low to Moderate Disease Activity. J Rheumatol. 2018 Aug;45(8):1078-1084. doi: 10.3899/jrheum.170770. Epub 2018 Apr 15. PMID 29657146

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Vanderbilt Rheumatology practice, responses to advertisements, and word of mouth. Exclusion criteria included estimated glomerular filtration rate of <60 ml/min and inability to undergo cardiac MRI.
Groups:
- Rheumatoid Arthritis Patients: People who have rheumatoid arthritis
- Controls: people who do not have RA or other inflammatory disease
Period: Overall Study
Arm/Group | Rheumatoid Arthritis Patients | Controls
Started | 67 | 61
Completed | 59 | 56
Not Completed | 8 | 5
Not completed — EGFR <60ml/min | 6 | 4
Not completed — claustrophobic when entering cardiac MRI | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rheumatoid Arthritis Patients | Controls | Total
Number analyzed (Participants) | 59 | 56 | 115
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 53 [40 to 59] | 52 [38 to 57] | 53 [38 to 59]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 44 | 89
  Male | 14 | 12 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 58 | 55 | 113
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 59 | 56 | 115

OUTCOME MEASURES:

1. Primary Outcome: Left Ventricular Mass Indexed to BSA, g/m^2
Description: Left Ventricular Mass (LVM) is known to increase in proportion to overall body size and differs by gender. To assess an individual's risk for a cardiovascular event based on LVM,an adjustment for the patient's body size should be done. LVM in grams was divided by body surface area in meters squared, to adjust for body size. Body surface area was calculated by square root (height (cm) X weight (kg)/3600).
Time Frame: one scan, cross sectional comparison
Measure: Median (Inter-Quartile Range); unit: g/m^2
Arm/Group | Rheumatoid Arthritis Patients | Controls
Number analyzed (Participants) | 59 | 56
g/m^2 | 43.8 [40 to 49.5] | 42.2 [36.4 to 48.5]

2. Secondary Outcome: Left Atrium Size, mm
Description: left atrium size, measured in millimeters
Time Frame: one scan, cross sectional comparison
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | Rheumatoid Arthritis Patients | Controls
Number analyzed (Participants) | 59 | 56
mm | 29 [24 to 32] | 29 [26 to 32]

ADVERSE EVENTS:
Time Frame: Research study was done in one day. Adverse events were recorded for the day that research study took place.
Arm/Group | Rheumatoid Arthritis Patients | Controls
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/61
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/61
Other Adverse Events (participants affected / at risk) | 0/67 | 0/61

LIMITATIONS AND CAVEATS:
Study is cross-sectional. Rheumatoid arthritis patients had low to moderate disease activity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No